CLINICAL TRIAL: NCT06836011
Title: Definition and Prognosis of Atrioventricular Regurgitation in Transthyretin Amyloid Cardiomyopathy - a Prospective International Multicenter Study
Brief Title: A Multicenter Study on Atrioventricular Regurgitation in Transthyretin Amyloid Cardiomyopathy: Definition, Prevalence, and Prognostic Impact.
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Nitsche, Priv.-Doz. Dr. med. univ., PhD, Medical University of Vienna
Other Study IDs: ATTR-CM-AVR-2025-001
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: ATTR Amyloidosis With Cardiomyopathy; ATTR-CM; ATTR Amyloidosis Wild Type; Mitral Regurgitation; Tricuspid Regurgitation
Keywords: ATTR-CM; ATTR amyloidosis; Tricuspid Regurgitation; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this prospective registry study is to comprehensively characterize the prevalence, (semi-) quantitative parameters, and associated clinical outcomes of mitral (MR) and tricuspid regurgitation (TR) in patients diagnosed with transthyretin amyloid cardiomyopathy (ATTR-CM). The study further aims to develop and implement new grading standards for the quantitative assessment of regurgitation severity, tailored to the distinct hemodynamic profile of ATTR-CM. This approach seeks to address the limitations of current regurgitation severity classifications, which do not adequately reflect the unique pathophysiology of a restrictive phenotype as seen in ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ATTR-CM according to current diagnostic criteria
* Comprehensive baseline echocardiographic assessment, including (semi-)quantitative mitral and tricuspid regurgitation (MR/TR) parameters, performed within ±6 months of diagnosis
* Age ≥ 18 years
* Willingness to participate in the study and provide informed consent

Exclusion Criteria:

* Severe aortic valve disease requiring intervention
* Inability to provide informed consent or participate in study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will include patients diagnosed with transthyretin amyloid cardiomyopathy (ATTR-CM) from international specialized cardiac amyloidosis referral centers. The study population will encompass both wild-type and hereditary ATTR-CM patients, ensuring representation of diverse disease phenotypes. Data collection will be standardized across centers, with echocardiographic assessments performed in accordance with the dedicated study protocol. The inclusion of multiple international centers will enhance the generalizability of findings across different healthcare systems and patient populations.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | up to 60 months
  Assessment of all-cause mortality in patients with ATTR-CM, stratified by baseline quantitative and semiquantitative measures of mitral and tricuspid regurgitation severity

SECONDARY OUTCOMES:
Cardiovscular mortality | up to 60 months
Heart Failure Hospitalization | up to 60 months
  Time to first heart failure hospitalization Rate of heart failure hospitalizations

OTHER OUTCOMES:
Progression of Atrioventricular Regurgitation | At 12 and 24 months follow-up
  Change in mitral and tricuspid regurgitation severity over time and its impact on clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (8):
- Austria (2):
  - Medical University of Graz, Graz, Styria
  - Department of Internal Medicine II, Medical University of Vienna, Vienna
- Germany (2):
  - Medizinische Klinik und Poliklinik I, Klinikum der Universitaet Muenchen, Ludwig-Maximilians-University, Munich, Bavaria
  - Department of Cardiology, University Hospital Frankfurt, Goethe University, Frankfurt am Main, Hesse
- Italy (3):
  - Institute of Cardiology, ASST Spedali Civili di Brescia, Department of Medical and Surgical Specialties, Radiological Sciences, and Public Health, University of Brescia, Brescia
  - Cardiologic Centre, Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Center for Diagnosis and Treatment of Cardiomyopathies, Cardiovascular Department, Azienda Sanitaria Universitaria Giuliano-Isontina (ASUGI), University of Trieste, Trieste
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dona C, Nitsche C, Koschutnik M, Heitzinger G, Mascherbauer K, Kammerlander AA, Dannenberg V, Halavina K, Rettl R, Duca F, Traub-Weidinger T, Puchinger J, Gunacker PC, Lamm G, Vock P, Lileg B, Philipp V, Staudenherz A, Calabretta R, Hacker M, Agis H, Bartko P, Hengstenberg C, Fontana M, Goliasch G, Mascherbauer J. Unveiling Cardiac Amyloidosis, its Characteristics, and Outcomes Among Patients With MR Undergoing Transcatheter Edge-to-Edge MV Repair. JACC Cardiovasc Interv. 2022 Sep 12;15(17):1748-1758. doi: 10.1016/j.jcin.2022.06.009. Epub 2022 Aug 22. PMID 36008266